## Title: Testing a Brief Substance Misuse Preventative Intervention for Parents/Guardians of 5th-7th Grade Students

NCT Number: NCT03925220

Informed Consent Form (Parents and Children-English and Spanish Versions)

Document Date: May 5, 2020

## TUFTS UNIVERSITY Department of Public Health and Community Medicine

#### INFORMED CONSENT TO PARTICIPATE IN RESEARCH

Principal Investigator: Margie R. Skeer, ScD, MPH, MSW Co-Investigators: Anthony Spirito, PhD; Misha Eliasziw, PhD

Study team telephone number: (617) 636-3587

#### INTRODUCTION

You are being invited to take part in a research study that is trying to understand how to help young people make choices that will support their well-being. Taking part in this research study is completely your choice. You can decide to stop at any time for any reason without any consequences.

Please read all of the following information carefully. Ask the research assistant to explain any words, terms, or sections that are unclear to you. Ask any questions that you have about this research study. Do not sign this consent form unless you understand the information in it and have had your questions answered.

If you decide to take part in this research study, you will be asked to sign this form. You will be given a copy of the signed form. You should keep your copy for your records. It has information, including important names and telephone numbers that you may want to look at in the future.

If you are able to participate and agree to be in the study, the Principal Investigator (the person who is in charge of the research study) may still choose to have you not be involved at some point during the study if she thinks it is best.

If you have any questions about your rights as a research study participant, call the Tufts Social-Behavioral-Educational Research IRB (Tufts SBER IRB): (617) 627-8804, <a href="mailto:sber@tufts.edu">sber@tufts.edu</a>. The Institutional Review Board is a group of doctors, nurses, and non-medical people who review research studies for safety and protection of people who take part in studies. Federal law requires the Institutional Review Board to review and approve any research study involving humans. This must be done before the study can begin. The study is also reviewed on a regular basis while it is in progress.

This research study has been reviewed and approved by the Tufts SBER IRB.

#### **PURPOSE OF STUDY**

The purpose of this study is to find out what parents like you can do to help children make choices that will support their well-being during their teenage years.

The National Institutes of Health is sponsoring this study. There are 500 parents/ children who attend public schools in the Greater Boston Area taking part in this study.

#### PROCEDURES TO BE FOLLOWED

If you take part in this study, it will last approximately 18 months, you will be chosen to be in one of two groups: Group A or Group B. Study participants will be chosen for Group A and Group B at random. Each group will be asked to complete a set of tasks, which are listed below.

- 1. Read a short book (called a handbook). After you finish reading this book, you will be asked to practice the skills you read about in the handbook.
- 2. Meet with an interventionist to go over what you read and complete an action plan. This meeting will give you a chance to ask any questions you have about what you read. It will most likely last about an hour. Within 2 weeks of this meeting, will also receive a brief follow-up phone call about what you discussed in the first meeting. Both sessions will be audio recorded.
- 3. Complete 5 surveys one at the beginning of the study, another 3, 6, 12, and 18 months after the study starts. Your child will also be asked to complete similar surveys at the same time
- 4. Video record four family meals at the beginning of the study and at 6- and 12-months.
- 5. Audio record one conversation you have about your child's well-being, as it pertains to this study, at baseline and at 3, 6,12, and 18 months. The study will provide you with an iPad to do the recordings, which will be yours to keep if you complete all recorded sessions over the entire study period. Your child will be recorded as part of the family meals and conversations.
- 6. Receive and read text messages that the research team will send to your cell phone or to a cell phone given to you for study purposes. The messages will be sent two times each week for 13 weeks. These text messages will have information from the handbook. You may also receive text messages to remind you about upcoming meetings or study tasks to complete. Your child will not get these text messages or any text messages from the research team.
- 7. At the start of the study, your child's height and weight will be taken.

Your child will only be asked to complete the surveys at the start of the study and at 3-, 6-, 12- and 18-months after the study starts and have their height and weight taken at the start of the study. He or she will not meet with the interventionist, will not be asked to read the handbook, and will not receive text messages as part of the study. Your child will be recorded as part of the family meals video recordings and the parent-child conversations.

Both you and your child have to agree to take part in this study. If one of you does not want to take part in the study then neither of you can be in the study. All of the meetings (surveys and meeting with the expert) will take place at your child's school, at your home, or at Tufts University School of Medicine located at 136 Harrison Ave, Boston MA (close to Chinatown in downtown Boston). However, if you are not able to meet at any of these places, the research assistant will work with you to find another place to meet that will be easy for you to get to. We may ask you to complete some surveys without meeting with a member of the study team. In this case, you will be contacted via phone, text message or email with instructions on how to complete the survey online.

#### **RISKS**

One potential risk of being in this study is that you may feel uncomfortable talking to the researcher about what you do with your child as a family. There is also a small chance that the

information you give us is given to someone else by accident. But we will do everything we can to make sure that this does not happen.

#### **BENEFITS**

This study will give you information that may help make your family a little stronger. It will also give you some things that you can do to help your child stay safe and healthy. Along with these individual benefits, the information you give us will also help others in society, particularly parents like you. This is because the information you provide the research team will allow us to create a larger program that works to help not only families living in the Greater Boston area, but families living in the United States.

#### **ALTERNATIVES**

The alternative is to not participate in the research study.

#### WHOM TO CONTACT

If you have any questions about this research study, you can call the Research Study Team (Tufts University) at (617) 636-3587; Dr. Margie R. Skeer, Principal Investigator (Tufts University): (617) 636-2441; or Dr. Anthony Spirito (Brown University): (401) 444-1929.

#### COSTS

You will have to get to and from the sessions and surveys that take place at your child's school, at Tufts University School of Medicine, or at the other location of your choosing. However, if you cannot get to an appointment, we can try to find a different place to meet.

#### **PAYMENT**

Your family will be paid \$60 in Amazon e-gift cards for completing each of the first, second, and third surveys, and \$80 in Amazon e-gift cards for completing each of the fourth and fifth surveys. Your family will be given payment after you both complete the survey.

### PRIVACY AND CONFIDENTIALITY

If you agree to take part in this research study, your personal information will not be given to anyone unless you tell us in writing that it is okay. The research team is made up of up of individuals from Tufts University and Brown University, which means your information will be shared among members of the research team at both schools when necessary. We will not share the information you give us with your child, and we will not share the information that your child gives us with you. We will try very hard to keep your information private. The National Institutes of Health, the Tufts SBER IRB, and the Grant Administration Office may check records that say who you are. This might include your research records and this informed consent form that you sign. The records of this study might also be looked at to make sure all rules and guidelines were followed. We, along with the Grant Administration Office that is in charge of study finances, will keep a copy of your signed payment acknowledgement form for our records.

In order to protect your privacy, all of your and your child's documents will be stored in locked cabinets. Documents for the study will have an ID number instead of your name and a document with your name and study ID number will be kept separately in a locked file. Any of your personal information, as well as this informed consent form, will be stored separately from your answers to questions that you write down on paper. Anything that we put on the computer will be stored and protected with a password and encrypted. Recordings will be reviewed by a study team member to make sure that nothing can identify you in the recordings. Once we have

written down the recordings they will be destroyed. Only the research team members will have access to the information in the recordings.

A description of this study will be posted on a public website, <a href="http://ClinicalTrials.gov">http://ClinicalTrials.gov</a> as required by our funding from the National Institutes of Health. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

Your data could be used for future research studies or shared with another investigator for future research purposes without additional informed consent from you or your legally authorized representative. In this event, all identifiers (any personal information identifying you) would be removed from the data set.

To help us protect your privacy, we have obtained a Certificate of Confidentiality from the United States Department of Health and Human Services (DHHS). With this Certificate, we cannot be forced (for example by court order or subpoena) to give information that may identify participants in any federal, state, local, civil, criminal, legislative, administrative, or other proceedings. Our research team will use the Certificate to resist any demands for information that would identify participants, except to prevent serious harm to participants or others.

However, if we learn about abuse of a child or elderly person, or that you intend to harm yourself or someone else, we will tell the proper authorities.

If your insurance company or job learns about your being in this study, and gets your permission to receive research information from us, then we may not use the Certificate of Confidentiality to hold back this information.

#### PARTICIPANT'S STATEMENT

I have read this consent form and have discussed the procedures described above with a member of the research team. I have been given the chance to ask questions, which have been answered as well as I want them to be. I understand that any questions that I might have will be answered through talking or, if I want, in writing.

I understand that I will be told about any new findings developed during the course of this research study that may change whether I want to stay in this research study.

I understand that I am in this study because I want to be. I understand that I may choose to stop being in this study. I also understand that if, for any reason, I want to stop being in this study at any time, I can, and this will not change how I can get services or care at any participating research site.

I understand that if I get sick or hurt from being in this research study, medical care will be given to me. However, this medical care will not be free, even if the sickness or injury is a direct result of this research study. I understand that no money is provided to pay for care if I get sick or hurt as part of this study.

If I have any questions concerning my rights as a research participant in this study, I may contact the Institutional Review Board at (617) 627-8804.

I have been fully told about the study with its risks and benefits, and I am willing to take part in the procedures for this study, as it talks about in this form.

I understand that as a participant in this study my personal information and data relating to this research study will be kept private, except as required by law, and except for inspections by the U.S. Food and Drug Administration, which regulates investigational drug/device studies, the study sponsor.

## By clicking "I agree to be part of the SUPPER Project Study" you agree to the following:

- I consent to participate in the study.
- I also provide consent for my child to participate in this study, as it talks about in this form.
- I will complete the survey myself without assistance from anyone except a research team member,
- I will not share my responses with my child; and
- I will not watch or help my child complete their survey.

I agree to be part of the SUPPER Project Study

# UNIVERSIDAD DE TUFTS Departamento de Salud Pública y Medicina Comunitaria

#### CONSENTIMIENTO INFORMADO PARA PARTICIPAR EN LA INVESTIGACIÓN

Investigadora Principal: Margie R. Skeer, ScD, MPH, MSW Co-Investigadores: Anthony Spirito, PhD, Misha Eliasziw, PhD Número telefónico del Equipo de Investigación: (617) 636-3587

### INTRODUCCIÓN

Usted ha sido invitado(a) a ser parte de un estudio que está tratando de entender cómo podemos ayudar a los jóvenes a tomar decisiones que les ayudará con su bienestar. Tomar parte en este estudio de investigación es completamente su decisión. Usted puede parar de participar en cualquier momento y por cualquier razón, sin ninguna consecuencia.

Por favor lea la siguiente información cuidadosamente. Pida al asistente de investigación que le explique cualquier palabra, término o sección que no esté clara para usted. Haga cualquier pregunta que tenga sobre este estudio de investigación. Sólo firme este consentimiento informado si ha entendido la información del mismo y cuando todas sus preguntas hayan sido respondidas.

Si usted decide formar parte de este estudio de investigación, le pediremos que firme esta forma. Le entregaremos una copia de la forma firmada para sus archivos. Usted deberá mantener una copia en sus archivos. Éstas tienen información que incluyen nombres y números telefónicos que usted pudiera querer utilizar en el futuro.

Si usted puede participar y acepta participar en el estudio; es posible que la Investigadora Principal (la persona responsable del estudio) pudiera decidir que usted no participe en cualquier momento del estudio si ella considera que sería para lo mejor.

Si usted tiene alguna pregunta sobre sus derechos como participante en un estudio de investigación, llame al Comité Institucional de Revisión para las investigaciones en las Ciencias Sociales, del Comportamiento y Educacionales de la Universidad de Tufts (Tufts SBER IRB): (617) 627-8804, sber@tufts.edu. El Comité Institucional de Revisión está compuesto por un grupo de doctores, enfermeras y personal no médico quienes revisan los estudios para garantizar la seguridad y protección de las personas que participan en los estudios. Las leyes federales requieren que el Comité Institucional de Revisión revise y apruebe cualquier estudio de investigación con seres humanos. Esto tiene que ser hecho antes de que el estudio comience. El estudio también es revisado regularmente mientras está tomando lugar.

Este estudio ha sido revisado y aprobado por el IRB de Tufts SBER.

#### PROPÓSITO DEL ESTUDIO

El propósito de este estudio es averiguar qué los padres como usted pueden hacer para ayudar a sus hijos(as) a tomar decisiones que los ayudarán con su bienestar en su adolescencia.

El Instituto Nacional de Salud está patrocinando este estudio. Hay 500 padres/niños que asisten a Escuelas Públicas en Boston y en las áreas alrededor de Boston tomando parte en este estudio.

#### PROCEDIMIENTO A SEGUIR

Si usted decide participar en este estudio, durará aproximadamente 18 meses, usted será elegido a uno de dos grupos: Grupo A o Grupo B. Los participantes del estudio serán elegidos al Grupo A y al Grupo B al azar. A cada grupo se les pedirá que completen una serie de tareas, que se enumeran a continuación.

- 1. Leer un libro corto (llamado manual). Después que termine de leer el libro, le pediremos que practique las destrezas que leyó en el libro.
- 2. Reunirse con un intervencionista para hablar sobre lo que usted leyó y completar un plan de acción. Esta reunión le dará la oportunidad de hacer cualquier pregunta que usted tenga sobre lo que leyó. Ésta reunión durará aproximadamente una hora. Esta sesión será audio grabada. Dentro de 2 semanas de esta reunión, usted también recibirá una breve llamada telefónica que le dará seguimiento a lo que discutieron en la primera reunión.
- 3. Completar cinco encuestas- una al inicio del estudio, a los 3, 6, 12, y 18 meses de empezar el programa. También se le pedirá a su hijo(a) que complete encuestas similares al mismo tiempo.
- 4. Vídeo grabar cuatro comidas en familia al inicio del estudio y a los 6 y 12 meses. Audio grabar una conversación que usted tenga acerca del bienestar de su hijo(a) relacionada con el estudio al principio del estudio y a los 3, 6, 12 y 18 meses. Las grabaciones se llevarán a cabo con un iPad que el estudio le proporcionará a usted, la cuál será suya si completa todas las grabaciones durante la duración del estudio. Su hijo(a) será parte de las grabaciones de las comidas en familia y las conversaciones.
- 5. Recibir y leer mensajes de texto que el equipo de investigación le enviará a su teléfono celular o al teléfono celular que será entregado para los propósitos del estudio. Estos mensajes serán enviados 2 veces por semana durante 13 semanas. Estos mensajes tendrán información de los manuales y también recordatorios acerca de futuras reuniones. Su hijo no recibirá ninguno de estos mensajes de texto ni ningún otro tipo de mensaje enviado por el equipo de investigación.
- 6. Al inicio del estudio, mediremos la altura y peso de su hijo(a).

A su hijo(a) sólo se le pedirá que complete las encuestas como parte del estudio y que se le mida su altura y peso al inicio del estudio. Él o ella no se reunirá con el intervencionista, no se le pedirá que lea el manual ni recibirá mensajes de texto como parte del estudio. Su hijo(a) será grabado como parte de las vídeo grabaciones de las comidas en familia.

Ambos usted como su hijo(a) deberán estar de acuerdo en participar en este estudio. Si uno de los dos no desea tomar parte en el estudio, ninguno de los dos podrá participar en el estudio. Todas las reuniones (las encuestas y la reunión con el experto) tomarán parte en la escuela del niño(a), en su hogar, o en la Escuela de Medicina de la Universidad de Tufts, que está ubicada en 136 Harrison Ave, Boston MA (cerca de Chinatown en el Centro de Boston). Sin embargo, si usted no puede reunirse en ninguno de estos lugares, el/la asistente de investigación le ayudará a encontrar otro lugar más conveniente para usted, donde podrán reunirse. Es posible que le pidamos que complete estas encuestas sin reunirse con un miembro de nuestro equipo

de investigación. En dado caso, lo/a contactaremos por teléfono, mensajes de texto o correo electrónico con instrucciones de cómo completar las encuestas en línea.

#### **RIESGOS**

Un riesgo potencial al ser parte de este estudio es que usted podría sentirse incómodo(a) hablando con el investigador sobre lo que usted hace con su hijo(a) como familia. También hay una pequeña posibilidad de que la información que usted nos ha dado se le dé a otra persona por accidente. Pero nosotros haremos todo lo que sea posible para evitar que esto suceda.

#### **BENEFICIOS**

Este estudio le dará información que podría ayudarlo(a) a hacer que su familia sea un poco más fuerte. También le proporcionará algunas maneras de cómo hablar con su hijo(a) sobre cosas que él o ella pueden hacer para mantenerse sanos y a salvo. Junto con estos beneficios individuales, la información que usted nos da también ayudará a otros en la sociedad, en particular a otros padres como usted. Esto se debe a que la información que usted le proporcionará al equipo de investigación nos permitirá crear un programa más amplio que ayudará no sólo a las familias que viven en Boston, sino también a las familias que viven en los Estados Unidos.

#### **ALTERNATIVAS**

La alternativa es no participar en el estudio de investigación.

## A QUIÉN CONTACTAR

Si usted tiene alguna pregunta sobre este estudio de investigación usted puede llamar a la administradora del proyecto, Rachael Sabelli (Universidad de Tufts) al (617) 636-3651; a la Dra. Margie R. Skeer, Investigatora Principal (Universidad de Tufts): (617) 636-2441; o al Dr. Anthony Spirito (Universidad de Brown): (401) 444-1929.

### COSTOS

Usted tendrá que ir y venir de las sesiones y encuestas que se llevan a cabo en la escuela de su hijo(a) o en la Escuela de Medicina de la Universidad de Tufts. De todas formas, si usted no puede llegar a una cita, nosotros podemos tratar de encontrar un lugar diferente para reunirnos.

#### **PAGO**

Le pagaremos a su familia \$60 en tarjetas de regalo electrónicas de Amazon por la primera, segunda y tercera encuesta (cada una), y \$80 en tarjetas de regalo electrónicas de Amazon por completar la cuarta y quinta encuesta (cada una). Su familia recibirá el pago cuando ambos completen la encuesta.

### PRIVACIDAD Y CONFIDENCIALIDAD

Si usted decide participar en este estudio de investigación, su información personal no se le entregará a nadie a no ser que usted nos diga por escrito, que podemos hacerlo. El equipo de investigación está compuesto por individuos de la Universidad de Tufts y de la Universidad de Brown; lo cual quiere decir, que su información será compartida entre miembros de las dos universidades cuando sea necesario. Nosotros no compartiremos la información que usted nos dé con su hijo(a) o la información que él/ella nos dé con usted. Haremos todo lo posible para mantener su información privada. El Instituto Nacional de Salud, el Comité Institucional de Revisión SBER Tufts, y la Oficina de Administración de Fondos podrían revisar archivos que digan quién es usted. Esto puede incluir sus archivos de la investigación y este consentimiento

informado con su firma. Los archivos de este estudio podrían ser revisados para asegurar que las reglas de este estudio sean cumplidas. Nosotros, con la Oficina de Administración de Fondos que se encarga de las finanzas del estudio, guardaremos una copia de su formulario firmado de recibo de pago para nuestros archivos.

Para proteger su privacidad, todos sus documentos y los de su hijo(a) serán guardados en un gabinete con llave. Los documentos del estudio tendrán un número de identificación en lugar de su nombre. Un documento con su nombre y número de identificación del estudio será archivado en un gabinete separado y con llave. Su información personal, así como el consentimiento informado serán guardados separados de sus respuestas a las preguntas que usted completó en papel. Cualquier información que pongamos en la computadora será guardada y protegida con una clave y encriptada. Las grabaciones serán revisadas por un miembro del equipo de investigación para asegurar que no haya nada que lo pueda identificar a usted. Cuando hayamos escrito las grabaciones, estás serán destruidas. Sólo los miembros del equipo de investigación tendrán acceso a la información de las grabaciones.

Una descripción del estudio será publicada en un sitio web público, <a href="http://ClinicalTrials.gov">http://ClinicalTrials.gov</a> como requisito de nuestra financiación del Instituto Nacional de Salud (NIH). Este sitio web no incluirá información que le pueda identificar. Como máximo, el sitio web incluirá un resumen de los resultados. Usted puede buscar este sitio web en cualquier momento.

Sus datos podrían ser usados para futuros estudios de investigación o compartidos con otro investigador para futuros propósitos de investigación sin consentimiento informado adicional de usted o su representante autorizado legal. En este evento, todos los identificadores (cualquier información personal identificándole) serán removidos del conjunto de datos.

Para ayudarnos a proteger su privacidad hemos obtenido un Certificado de Confidencialidad del Departamento de Servicios Humanos y Salud (DHHS) de los Estados Unidos. Con este certificado, nosotros no podemos ser forzados (ejemplo: por una orden de la corte o citación) a dar información que pueda identificar participantes en ningún procedimiento federal, estatal, local, civil, criminal, legislativo, administrativas o de otro tipo. Nuestro equipo de investigación usará este Certificado para resistir cualquier demanda de información que pudiera identificar participantes con la excepción de prevenir daños serios a participantes u otras personas.

Sin embargo, si sabemos sobre el abuso de un niño o una persona de edad avanzada o que tiene la intención de hacerse daño a sí mismo(a) o a otra persona, se lo reportaremos a las autoridades apropiadas.

Si su compañía de seguro o trabajo sabe sobre su participación en este estudio y recibe su permiso para obtener información de nuestra investigación, entonces nosotros no usaremos el Certificado de Confidencialidad para retener esa información.

## **DECLARACIÓN DEL PARTICIPANTE**

Yo he leído este consentimiento informado y he discutido los procedimientos descritos anteriormente con un miembro del equipo de investigación. He tenido la oportunidad de hacer preguntas, las cuales han sido contestadas tan bien como yo quisiera. Yo entiendo que cualquier otra pregunta que yo pudiera tener será respondida verbalmente o si yo quisiera, por escrito.

Yo entiendo que me dirán sobre cualquier nuevo descubrimiento desarrollado durante el curso de este

estudio de investigación que pudiera cambiar el que yo quiera continuar participando en el estudio.

Yo entiendo que yo estoy en el estudio porque yo quiero estarlo. Yo entiendo que puedo decidir dejar de participar en el estudio. Yo también entiendo que si por alguna razón quiero dejar de participar en este estudio, en cualquier momento, yo puedo y esto no cambiará la forma en la que recibo servicios o cuidados en cualquiera de los sitios que están participando en este estudio.

Yo entiendo que si me enfermo o me lesiono por estar en este estudio de investigación, recibiré cuidados médicos. Sin embargo, estos cuidados médicos no serán gratuitos, aún si la enfermedad o lesión es consecuencia directa de este estudio de investigación. Yo entiendo que ninguna cantidad de dinero será entregada para pagar por cuidados si yo me enfermo o lesiono como parte de este estudio.

Si tengo preguntas relacionadas con mis derechos como participante en este estudio yo puedo contactar al Comité Institucional de Revisión llamando al (617) 627-8804.

Yo he sido completamente informado(a) sobre el estudio con sus riesgos y beneficios y estoy dispuesto(a) a ser parte de los procedimientos de este estudio como se han explicado en esta forma.

Yo entiendo que como participante en este estudio mi información personal y datos relacionados con este estudio serán mantenidos en privado, a excepción de lo requerido por la ley y excepto a las inspecciones del Departamento de Drogas y Alimentos de los Estados Unidos, el cuál regula investigaciones de medicamentos/dispositivos, el patrocinador del estudio.

## Al hacer clic en "Yo estoy de acuerdo en ser parte del Proyecto SUPPER" usted está de acuerdo con lo siguiente:

- Doy consentimiento a participar en este estudio
- Doy consentimiento a mi hijo(a), como se describe en este formulario
- Yo completaré la encuesta por mí mismo(a) sin la asistencia de nadie excepto de un miembro del estudio
- No compartiré mis respuestas con mi hijo(a), y
- No miraré ni ayudaré a mi hijo(a) a completar su encuesta

Yo estoy de acuerdo en ser parte del Proyecto SUPPER

## TUFTS UNIVERSITY Department of Public Health and Community Medicine

#### AGREEMENT TO PARTICIPATE IN RESEARCH

Principal Investigator: Margie R. Skeer, ScD, MPH, MSW Co-Investigators: Anthony Spirito, PhD; Misha Eliasziw, PhD

We are asking you to take part in a research study we are doing. A research study is a way to learn about something in medicine and/or health. For this study, we would like to find out more about what family practices make pre-teens and teenagers more or less likely to do things that keep them safe and healthy.

We are asking you to be in the study because we think you will give us really important information about why children do things that support their overall well-being.

If you agree to take part this study, we will ask you to complete 5 surveys that will each last about an hour - one at the beginning of the study, another 3, 6, 12, and 18 months after the program starts. You will complete these surveys on a computer or tablet. You can complete these surveys at your school, at Tufts University in Boston, at your home, or at another place that your parent or guardian chooses. You will meet with a research team member to show you how to complete the surveys online by yourself, after that you may be asked to complete them while meeting with a study team member, or online. The questions on the survey will ask you about your family practices and what you do at home, as well as your thoughts and how often you take part in different behaviors that can help you stay safe and healthy. The survey will take place without your parent or guardian there. Your parent or guardian will also complete a survey about your family practices, but we will not share with your parent or guardian's survey answers with you.

At the beginning of the study, we will also take your height and weight measurements. Your measurements will be kept private and will only be used for study purposes.

We will also ask that your parent/guardian video record four family meals at the beginning of the study and at 6- and 12-months. We will also ask that your parent/guardian video or audio record one conversation you have about behaviors that support your well-being at each study visit at the beginning of the study and at 3, 6, 12 and 18 months. Recordings will be done using a tablet that will be provided to your family by the study, which will be your family's to keep if all recordings over the entire study period are completed. You and your parent/guardian will both be included in all the recordings.

We hope that by taking part in this study, you will help us learn some things that could help us figure out how to help teenagers make choices that will keep them safe and healthy.

You may feel uncomfortable talking about yourself or your family. If you do at any time, you can stop answering the questions. You do not have to be part of this study. It is up to you. You can say yes now and change your mind later. All you have to do is tell us that you want to stop. We will not be mad at you if you do not want to be in the study. We will not be mad if you join the study now and change your mind later.

If you have any questions about this research study, you can call the Research Study Team (Tufts University) at (617) 636-3587; Dr. Margie R. Skeer, Principal Investigator (Tufts University): (617) 636-2441; or Dr. Anthony Spirito (Brown University): (401) 444-1929.

A description of this study will be posted on a public website, <a href="http://ClinicalTrials.gov">http://ClinicalTrials.gov</a> as required by our funding from the government. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

Your data could be used for future research studies or shared with another researcher for future research purposes without additional assent from you or additional consent from your parent or legally authorized representative. In this event, any personal information identifying you would be removed from the data set.

To help us protect you, we have a certificate from the government, called a Certificate of Confidentiality. With this certificate, we cannot be forced to give your information to anyone. But, if at any time you tell someone on the research team that you are being hurt or abused by someone, we will tell the proper authorities, meaning the police or other officials.

Before you say yes or no to being in this study, you can ask us any questions. You can ask questions about the study at any time. Just tell me or anyone else on the research staff that you have a question.

Your family will get \$60 for each of the first three surveys completed and \$80 for each of the last two surveys completed.

By clicking "I agree to be part of the SUPPER Project Study" you agree to participate in the SUPPER Project.

I agree to be part of the SUPPER Project Study

## UNIVERSIDAD DE TUFTS Departamento de Salud Pública y Medicina Comunitaria

### ACUERDO PARA PARTICIPAR EN EL ESTUDIO DEINVESTIGACIÓN

Investigadora Principal: Margie R. Skeer, ScD, MPH, MSW Co-Investigadores: Anthony Spirito, PhD;

Misha Eliasziw, PhD

Te estamos pidiendo que participes en un estudio de investigación que estamos haciendo. Un estudio de investigación es una manera de aprender algo en la medicina y/o acerca de la salud. Para este estudio, nos gustaría averiguar más acerca de cuáles costumbres en familia hacen que sea más o menos probable que los pre-adolescentes y adolescentes hagan cosas que los mantengan sanos y a salvo.

Te estamos pidiendo que participes en el estudio porque pensamos que nos podrías dar información muy importante acerca del porqué los niños hacen cosas que les ayudan con su bienestar en general.

Si estás de acuerdo en participar en este estudio, te pediremos que completes 5 encuestas que tomarán como una hora cada una- una al inicio del estudio, otra a los 3, 6, 12 y 18 meses después que el programa empiece. Completarás estas encuestas en la computadora o en una tableta. Puedes completar estas encuestas en tu escuela, en la Universidad de Tufts en Boston, en tu hogar, o en cualquier otro lugar donde tu padre/encargado escoja. Te reunirás con un miembro del estudio para mostrarte como completar las encuestas en línea por ti mismo(a), después se te pedirá que las completes cuando te vuelvas a reunir con un miembro del estudio o en línea. Las preguntas en la encuesta te preguntarán acerca de costumbres en tu familia y lo que haces en casa, y también lo que piensas y cada cuánto tomas parte en diferentes conductas que te ayudan a mantenerte sano(a) y a salvo. Las encuestas se harán sin que esté tu padre o encargado presente. Tu padre o encargado también completará una encuesta acerca de las costumbres en tu familia, pero no compartiremos con tu padre o encargado lo que tú escribas en tu encuesta. Tampoco compartiremos contigo lo que tu padre o encargado ha escrito en su encuesta.

Al inicio del estudio, también tomaremos medidas de tu altura y peso. Tus medidas se mantendrán confidenciales y serán usadas solamente para el estudio.

También le pediremos a tu padre o encargado que grabe vídeos de cuatro comidas familiares al inicio del estudio y a los 6 y 12 meses. También le pediremos a tu padre o encargado que grabe videos o audios de una conversación que ustedes tengan acerca de conductas que le ayudan a tu bienestar en cada visita del estudio, al inicio del estudio, a los 3, 6, 12 y 18 meses. Las grabaciones se harán con una tableta que el estudio le dará a tu familia, que podrá ser de ustedes si completan todas las grabaciones durante el estudio. Tú y tu padre o encargado aparecerán en todas las grabaciones.

Esperamos que, al tomar parte en este estudio, tú nos ayudarás a aprender algunas cosas que nos ayudarán a averiguar cómo podemos ayudar a los adolescentes a tomar decisiones que los ayudarán a mantenerse sanos y a salvo.

Puede que te sientas incomodo(a) al hablar acerca de ti o de tu familia. Si te sientes así en algún momento, puedes parar de responder a las preguntas. No tienes que tomar parte en este estudio. Es tu decisión. Puedes decir que sí ahora y cambiar de opinión luego. Lo único que tienes que hacer es

decirnos que quieres parar de participar. No nos enojaremos contigo si no quieres ser parte del estudio. No nos enojaremos si te unes al estudio ahora y luego cambias de opinión.

Si tienes alguna pregunta acerca del estudio, puedes llamar al equipo de estudio de investigación (Universidad de Tufts) al (617) 636-3587; Dr. Margie R. Skeer, Investigadora Principal (Universidad de Tufts): (617) 636-2441; o Dr. Anthony Spirito (Universidad de Brown): (401) 444-1929.

Una descripción del estudio será publicada en un sitio web público, <a href="http://ClinicalTrials.gov">http://ClinicalTrials.gov</a> como requisito de nuestra financiación del gobierno. Este sitio web no incluirá información que te pueda identificar. Como máximo, el sitio web incluirá un resumen de los resultados. Tú puedes buscar este sitio web en cualquier momento.

Tus datos podrían ser usados para futuros estudios de investigación o compartidos con otro investigador para futuros propósitos de investigación sin asentimiento adicional tuyo o consentimiento de tu padre o representante autorizado legal. En este evento, cualquier información personal identificándote serán removidos del conjunto de datos.

Para ayudarnos a protegerte, tenemos un certificado del gobierno que se llama Certificado de Confidencialidad. Con este certificado, nadie nos puede obligar a darle tu información a nadie. Pero, si en algún momento tú le dices a un miembro del estudio que alguien te lastima o te abusa, nosotros le podemos decir a las autoridades apropiadas, es decir, a la policía ú otros oficiales.

Antes que digas que sí o no al estudio, nos puedes preguntar cualquier pregunta. Nos puedes preguntar acerca del estudio en cualquier momento. Sólo me tienes que decir a mí o a cualquier otro miembro de la investigación que tienes una pregunta.

Si firmas tu nombre abajo, significa que estás de acuerdo en tomar parte en este estudio. Tu familia recibirá \$60 por cada una de las tres encuestas completadas y \$80 por cada una de las dos últimas encuestas completadas.

Al hacer clic en "Yo estoy de acuerdo en ser parte del Proyecto SUPPER" tú estás de acuerdo en participar en el Proyecto SUPPER.

Yo estoy de acuerdo en ser parte del Proyecto SUPPER